CLINICAL TRIAL: NCT06800924
Title: Analysis of Posture and Spinal Mobility in Women Suffering From Anorexia Nervosa
Brief Title: Posture and Spinal Mobility in Anorexia Nervosa
Acronym: SPINALAN
Status: Active, not recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 01C416
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa; Spinal mobility; Posture
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anorexia Nervosa: Women suffering from anorexia nervosa clinically diagnosed based on the DSM-5 criteria (Diagnostic and Statistical Manual of Mental Disorders 5; American Psychiatric Association, 2013), aged ≥ 18 years
  Interventions: Other: Postural and mobility analysis
- Normal weight: Normal-weight adult women (age: ≥ 18 years; BMI: 18.5-24.9 kg/m2), recruited from the medical/nursing and research staff.
  Interventions: Other: Postural and mobility analysis

INTERVENTIONS:
Other: Postural and mobility analysis — Postural and mobility parameters were obtained with the use of the Idiag M360 scan tool (Idiag, Fehraltorf, Switzerland)

SUMMARY:
The primary objective of the study is to compare the results of the postural and mobility analysis obtained with the use of the Idiag M360 instrument in adult women with anorexia nervosa and in a control group represented by age-matched normal-weight women.

Secondary objectives will be to correlate the results obtained from previous postural analyses with anthropometric parameters, the duration and onset of the disease, and the presence/date of onset of secondary amenorrhea.

ELIGIBILITY:
Anorexia Nervosa:

Inclusion Criteria:

* Female sex
* Age 18 years and older
* Anorexia nervosa clinically diagnosed based on the DSM-5 criteria
* Hospitalized in the Division of Eating and Nutrition Disorders (END), Istituto Auxologico Italiano, IRCCS, Piancavallo (VB), Italy

Exclusion Criteria:

* Absence of signed informed consent
* Musculoskeletal or neurological conditions (leg length discrepancy, spinal deformities, and physical disabilities caused by surgery)
* Treatment with anti-inflammatory drugs

Normal Weight:

Inclusion Criteria:

* Female sex
* Age 18 years and older
* BMI: 18.5-24.9 kg/m2
* Recruited from the medical/nursing and research staff

Exclusion Criteria:

* Absence of signed informed consent
* Musculoskeletal or neurological conditions (leg length discrepancy, spinal deformities, and physical disabilities caused by surgery)
* Treatment with anti-inflammatory drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects admitted to the study will be recruited at the beginning of hospitalization in the Division of Eating and Nutrition Disorders (END), Istituto Auxologico Italiano, IRCCS, Piancavallo (VB), Italy. Thirty women suffering from anorexia nervosa clinically diagnosed based on the DSM-5 criteria (Diagnostic and Statistical Manual of Mental Disorders 5; American Psychiatric Association, 2013), aged ≥ 18 years, will be studied.
  As a control group, 30 normal-weight adult women (age: ≥ 18 years; BMI: 18.5-24.9 kg/m2) will be recruited from the medical/nursing and research staff.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Lateral flexion | Baseline
  Idiag M360 scan tool (Idiag, Fehraltorf, Switzerland); flexion expressed in degrees
Lumbar flexion | Baseline
  IIdiag M360 scan tool (Idiag, Fehraltorf, Switzerland); flexion expressed in degrees
Lumbar extension | Baseline
  IIdiag M360 scan tool (Idiag, Fehraltorf, Switzerland); extension expressed in degrees
Thoracic extension | Baseline
  IIdiag M360 scan tool (Idiag, Fehraltorf, Switzerland); extension expressed in degrees

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Site Piancavallo, Oggebbio, Verbania, Italy